CLINICAL TRIAL: NCT00422162
Title: An Eight-Week, Randomized, Double Blind, Two Parallel Groups, Study to Assess Clinical Response of Duloxetine 60 mg and 120 Per Day in Patients Hospitalized for Severe Depression
Brief Title: A Study Evaluating Duloxetine in Patients Hospitalized for Severe Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10614; F1J-BI-HMES (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Duloxetine Hydrochloride (60 mg) (Experimental): Up to Week 4: 60 milligrams (mg) every morning and placebo every evening, by mouth (PO).
  Week 4 to Week 8: Responders continued on same dose as before; Nonresponders received 60 mg every morning and 60 mg every evening added to the placebo
  Interventions: Drug: Duloxetine hydrochloride; Drug: Placebo
- Duloxetine Hydrochloride (120 mg) (Experimental): Up to Week 4: 60 mg every morning and 60 mg every evening, PO.
  Week 4 to Week 8: Responders continued on same dose as before; Nonresponders continued as before with a placebo capsule added to the evening dose
  Interventions: Drug: Duloxetine hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine hydrochloride — 60 mg once or twice a day, by mouth
  Other Names: LY248686; Cymbalta
Drug: Placebo — placebo capsule by mouth

SUMMARY:
An eight-week, randomized, double blind, two parallel groups, study to assess clinical response of duloxetine 60 milligrams (mg) and 120 mg per day in patients hospitalized for severe depression.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients of ≥ 18 years of age that meet criteria for severe Major Depressive Disorder, without psychotic features (according to Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, [DSM-IV] and confirmed by Mini International Neuropsychiatric Interview [MINI]).

* With a total score Montgomery-Asberg Depression Rating Scale (MADRS) ≥ 30 and 6-item Hamilton Depression Rating Scale (HAMD-6) ≥ 12 and Clinical Global Impression of Severity (CGI-Severity) ≥ 4 at both screening and baseline.
* Requirement of hospitalization (not for social or other non-medical reasons) at screening visit and at least up to Visit 4.
* Patients willing and able to comply with the requirement for hospitalization and with all scheduled visits, tests and procedures required by the protocol.
* Informed consent document must be signed at screening visit, in accordance with Good Clinical Practice (GCP) and local regulatory requirements, prior to any study procedure.

Exclusion Criteria:

* More than two previous episodes of major depression that did not respond (according to investigator's opinion) to adequate doses and duration of two different antidepressant therapies.
* Lack of response to at least two antidepressant therapies given at adequate doses for at least 6 weeks for the current depressive episode.
* Concurrent presence of symptoms fulfilling criteria for any Axis I disorder other than anxiety disorders (with exception of the Obsessive-Compulsive Disorder (OCD)) or Major Depressive Disorder, in the investigator's judgment.
* Any previous diagnosis of a bipolar disorder, schizophrenia or OCD.
* Depression with catatonic features (according to DSM-IV), depression with post-partum onset, or organic mental disorders.
* The presence of an Axis II disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- France (17):
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Besançon
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Bordeaux
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Bully-les-Mines
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Château-Gontier
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Dijon
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Dole
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Fains-Véel
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Jarnac
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, La Charité-sur-Loire
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, La Rochelle
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Limoges
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Marseille
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Montberon
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Montpellier
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Nîmes
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Paris
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Saint-Dizier
- Italy (7):
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Florence
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Foggia
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Messina
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Milan
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Pisa
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Roma
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Siena
- Russia (6):
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Kazan'
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Lipetsk
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Moscow
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Nizhny Novgorod
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Saint Petersburg
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Saratov
- South Africa (5):
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Bryanston
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Cape Town
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, George
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Krugersdorp
  - For additional information regarding investigative sites for this trial contact 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559), Mon-Fri, 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST) or speak with your personal physician, Pretoria

REFERENCES:
- [Result] Brecht S, Desaiah D, Marechal ES, Santini AM, Podhorna J, Guelfi JD. Efficacy and safety of duloxetine 60 mg and 120 mg daily in patients hospitalized for severe depression: a double-blind randomized trial. J Clin Psychiatry. 2011 Aug;72(8):1086-94. doi: 10.4088/JCP.09m05723blu. Epub 2010 Sep 21. PMID 20868642
- [Derived] Demyttenaere K, Desaiah D, Raskin J, Cairns V, Brecht S. Suicidal thoughts and reasons for living in hospitalized patients with severe depression: post-hoc analyses of a double-blind randomized trial of duloxetine. Prim Care Companion CNS Disord. 2014;16(3):PCC.13m01591. doi: 10.4088/PCC.13m01591. Epub 2014 May 1. PMID 25317365
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 392 patients who signed informed consent, 339 were randomized.
Groups:
- Duloxetine (60 mg): 60mg every day (QD) for 4 weeks, then responders continued on same dose and nonresponders increased to 60mg twice a day (BID) for next 4 weeks
- Duloxetine (120 mg): 60mg BID for 8 weeks (placebo added at Week 4 for nonresponders)
Period: Overall Study
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Started | 167 | 172
Received Treatment | 167 | 171
Completed | 143 | 142
Not Completed | 24 | 30
Not completed — Adverse Event | 11 | 9
Not completed — Lack of Efficacy | 4 | 10
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Non-Compliant with Protocol | 1 | 1
Not completed — Other | 0 | 1
Not completed — Didn't Receive Treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg) | Total
Number analyzed (Participants) | 167 | 171 | 338
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.9) | 43.9 (12.7) | 44.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 133 | 251
  Male | 49 | 38 | 87
Region of Enrollment [Number; unit: participants]
  France | 64 | 64 | 128
  South Africa | 15 | 17 | 32
  Russian Federation | 81 | 84 | 165
  Italy | 7 | 6 | 13
Previous Major Depressive Disorder Episodes [Number; unit: participants]
  Yes | 144 | 150 | 294
  No | 23 | 21 | 44
Race/Ethnicity [Number; unit: participants]
  Asian | 2 | 0 | 2
  Black | 4 | 8 | 12
  Caucasian | 161 | 163 | 324
Age at First Major Depressive Episode [Mean (Standard Deviation); unit: years] | 36.3 (13.3) | 35.6 (12.4) | 36.0 (12.8)
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic Blood Pressure | 118.7 (12.4) | 119.4 (14.8) | 119.1 (13.7)
  Diastolic Blood Pressure | 74.6 (8.5) | 74.7 (8.2) | 74.7 (8.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight in kilograms divided by height in meters squared.
  kilograms/square meter (kg/m^2) | 25.2 (5.5) | 25.5 (5.5) | 25.3 (5.5)
Duration of Previous Major Depressive Disorder (MDD) Episode [Mean (Standard Deviation); unit: weeks] — Duration of previous MDD episode in participants who experienced a previous MDD episode.
  weeks | 16.4 (19.0) | 13.7 (11.3) | 15.0 (15.6)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 167.1 (8.1) | 166.5 (7.6) | 166.8 (7.9)
Number of Previous Hospitalizations [Mean (Standard Deviation); unit: number of hospitalizations] — Number of hospitalizations for MDD in participants who experienced previous MDD episodes.
  number of hospitalizations | 1.3 (1.6) | 1.5 (2.3) | 1.4 (2.0)
Number of Previous Major Depressive Disorder (MDD) Episodes [Mean (Standard Deviation); unit: number of episodes] — Number of previous MDD episodes for participants who experienced previous MDD episodes.
  number of episodes | 3.2 (2.7) | 3.1 (3.0) | 3.2 (2.9)
Pulse Rate [Mean (Standard Deviation); unit: beats per minute] | 76.0 (8.8) | 75.8 (9.2) | 75.9 (9.0)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 70.4 (16.7) | 70.6 (15.2) | 70.5 (15.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Week Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline to Week 4
Population: All randomized participants who received at least one dose of study drug; had baseline and at least one post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
units on a scale
  Baseline | 36.1 (4.0) | 36.0 (4.6)
  Change from Baseline | -20.1 (10.6) | -19.9 (10.0)
Statistical Analysis 1: Comparison: Duloxetine (60 mg) vs Duloxetine (120 mg); Test type: Superiority or Other; p = 0.88, ANCOVA — P-value for Change from Baseline. A priori alpha threshold was 0.05 with no adjustment for multiple testing; ANCOVA with stratification factors (country and pretreatment for MDD) and MADRS baseline as covariates and treatment regimen as the main factor

2. Secondary Outcome: Change in 6-Item Hamilton Depression Scale (HAMD-6) Total Scores From Baseline
Description: The HAMD-6 (Items 1,2,7,8,10,13 from the 17-item HAMD) evaluates "core" symptoms of Major Depressive Disorder (MDD). Total scores range from 0 (normal) to 22 (severe).
Time Frame: Baseline to Weeks 1, 2, 3, 4, 6, 8
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline value. Last observation carried forward. Participants were assigned their responder status at Week 4 and the data were retrospectively divided into these groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine 60 mg Responder: 60mg QD for 8 weeks
- Duloxetine 60 mg Non-Responder: 60mg QD for 4 weeks then 60mg BID for 4 weeks
- Duloxetine 120 mg Responder: 60mg BID for 8 weeks
- Duloxetine 120 mg Non-Responder: 60mg BID for 8 weeks (placebo added at Week 4)
- Duloxetine 60 mg (All): 60mg every day (QD) for 4 weeks, then responders continued on same dose and nonresponders increased to 60mg twice a day (BID) for next 4 weeks
- Duloxetine 120 mg (All): 60mg BID for 8 weeks (placebo added at Week 4 for nonresponders)
Arm/Group | Duloxetine 60 mg Responder | Duloxetine 60 mg Non-Responder | Duloxetine 120 mg Responder | Duloxetine 120 mg Non-Responder | Duloxetine 60 mg (All) | Duloxetine 120 mg (All)
Number analyzed (Participants) | 96 | 70 | 106 | 64 | 166 | 170
units on a scale
  Change in Score at Week 1 | -3.9 (3.7) | -1.9 (3.2) | -3.3 (3.4) | -1.7 (2.7) | -3.1 (3.6) | -2.7 (3.3)
  Change in Score at Week 2 | -7.5 (4.4) | -3.4 (3.6) | -6.5 (4.2) | -3.0 (3.1) | -5.8 (4.6) | -5.2 (4.2)
  Change in Score at Week 3 | -9.4 (3.7) | -4.1 (3.4) | -8.7 (3.6) | -3.6 (3.7) | -7.2 (4.4) | -6.8 (4.4)
  Change in Score at Week 4 | -11.0 (3.2) | -3.9 (3.3) | -10.7 (3.0) | -3.8 (3.6) | -8.0 (4.8) | -8.1 (4.7)
  Change in Score at Week 6 | -11.6 (3.5) | -6.4 (4.4) | -11.8 (3.3) | -5.5 (4.4) | -9.4 (4.7) | -9.4 (4.8)
  Change in Score at Week 8 | -12.3 (3.4) | -7.6 (5.1) | -12.5 (3.0) | -6.7 (5.4) | -10.3 (4.8) | -10.3 (4.9)

3. Secondary Outcome: Change in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score From Baseline
Description: as for outcome 1
Time Frame: Baseline to Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg Responder | Duloxetine 60 mg Non-Responder | Duloxetine 120 mg Responder | Duloxetine 120 mg Non-Responder | Duloxetine 60 mg (All) | Duloxetine 120 mg (All)
Number analyzed (Participants) | 96 | 70 | 106 | 64 | 166 | 170
units on a scale
  Change in Score at Week 1 | -10.3 (8.6) | -5.6 (6.2) | -8.8 (7.6) | -5.6 (6.3) | -8.3 (8.0) | -7.6 (7.3)
  Change in Score at Week 2 | -18.7 (9.9) | -9.4 (7.1) | -16.3 (8.4) | -8.9 (7.7) | -14.7 (9.9) | -13.5 (8.9)
  Change in Score at Week 3 | -23.2 (8.4) | -11.1 (6.8) | -20.9 (6.9) | -10.3 (9.1) | -18.1 (9.8) | -16.9 (9.3)
  Change in Score at Week 4 | -27.2 (6.5) | -10.4 (6.9) | -25.5 (5.6) | -10.5 (8.6) | -20.1 (10.6) | -19.9 (10.0)
  Change in Score at Week 6 | -28.3 (7.9) | -16.1 (9.4) | -28.1 (6.6) | -14.8 (10.4) | -23.1 (10.4) | -23.1 (10.5)
  Change in Score at Week 8 | -29.8 (7.3) | -19.0 (11.8) | -29.5 (6.6) | -17.2 (12.3) | -25.2 (10.8) | -24.9 (10.9)

4. Secondary Outcome: Evaluation of Rescue Options Based on Changes in the Montgomery-Asberg Depression Rating Scale (MADRS) and the 6-Item Hamilton Depression Scale (HAMD-6)
Description: Changes in Montgomery-Åsberg Depression Rating Scale (MADRS) and 6-Item Hamilton Depression Scale (HAMD-6) total scores were evaluated following dose up-titration in those patients who did not achieve the minimum 50% response for primary endpoint. MADRS is a rating scale for severity of depressive mood symptoms. Total scores range from 0 (low severity of symptoms) to 60 (high severity of symptoms). The HAMD-6, derived by the sum of HAMD-17 items 1, 2, 7, 8, 10 and 13, evaluates "core" symptoms of Major Depressive Disorder (MDD). Total subscale scores range from 0 (normal) to 22 (severe).
Time Frame: 4 to 8 weeks
Population: All randomized participants who received at least one dose of study drug and had a Week 4 and at least one following value. Last observation carried forward. Participants were assigned their responder status at Week 4 and the data were retrospectively divided into these groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg Responder | Duloxetine 60 mg Non-Responder | Duloxetine 120 mg Responder | Duloxetine 120 mg Non-Responder
Number analyzed (Participants) | 96 | 55 | 106 | 48
units on a scale
  Change in MADRS Score from Week 4 to Week 6 | -1.0 (5.1) | -7.2 (6.3) | -2.6 (4.2) | -5.8 (7.0)
  Change in MADRS Score from Week 4 to Week 8 | -2.6 (6.0) | -10.9 (8.8) | -4.0 (5.3) | -8.9 (9.1)
  Change in HAMD-6 Score from Week 4 to Week 6 | -0.6 (2.7) | -3.2 (2.7) | -1.1 (1.8) | -2.2 (3.1)
  Change in HMAD-6 Score from Week 4 to Week 8 | -1.3 (2.8) | -4.7 (3.6) | -1.8 (2.4) | -3.8 (4.3)

5. Secondary Outcome: Clinical Global Impression of Severity (CGI-S) Scores at Each Visit
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
units on a scale
  Week 0 (Baseline) | 5.0 (0.7) | 5.1 (0.7)
  Week 1 | 4.4 (0.9) | 4.4 (0.9)
  Week 2 | 3.6 (1.2) | 3.8 (1.1)
  Week 3 | 3.2 (1.3) | 3.4 (1.2)
  Week 4 | 3.0 (1.4) | 3.1 (1.3)
  Week 6 | 2.7 (1.4) | 2.7 (1.4)
  Week 8 | 2.3 (1.4) | 2.4 (1.5)

6. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Each Visit
Description: Measures clinician's perception of patient improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much better) to 7 (very much worse).
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
units on a scale
  Week 1 | 3.1 (0.8) | 3.2 (0.8)
  Week 2 | 2.5 (1.0) | 2.6 (0.8)
  Week 3 | 2.3 (0.9) | 2.3 (0.9)
  Week 4 | 2.3 (1.1) | 2.1 (1.0)
  Week 6 | 2.0 (1.1) | 2.0 (1.1)
  Week 8 | 1.9 (1.2) | 1.9 (1.1)

7. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Score at Each Visit
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Weeks 1, 2, 3, 4, 6, 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
units on a scale
  Week 1 (n=164, n=170) | 3.0 (1.0) | 3.1 (0.9)
  Week 2 (n=164, n=170) | 2.6 (1.1) | 2.6 (0.9)
  Week 3 (n=165, n=170) | 2.3 (1.1) | 2.4 (1.1)
  Week 4 (n=165, n=170) | 2.3 (1.2) | 2.2 (1.2)
  Week 6 (n=165, n=170) | 2.1 (1.3) | 2.0 (1.1)
  Week 8 (n=165, n=170) | 2.0 (1.3) | 1.9 (1.2)

8. Secondary Outcome: Hamilton Anxiety Scale (HAMA) Score at Baseline and Weeks 4 and 8
Description: The HAMA scale measures anxiety symptoms accompanying Major Depressive Disorder (MDD). Each item of the 14-item HAMA was scored from 0 (not present) to 4 (very severe), with a resulting maximum total score of 56.
Time Frame: Baseline and Weeks 4 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
units on a scale
  Week 0 (Baseline) (n=166, n=170) | 26.0 (6.4) | 27.0 (7.0)
  Week 4 (n=165, n=168) | 13.0 (8.8) | 13.4 (8.9)
  Week 8 (n=165, n=168) | 9.6 (8.8) | 9.8 (9.2)

9. Secondary Outcome: Percentage of Responders
Description: Patients with reduction in MADRS score ≥50% after 4 weeks were to stay on previous dose of duloxetine. Those with reduction in MADRS <50% were to receive 120 mg for remaining 4 weeks of treatment (up-titration from 60 mg to 120 mg for those randomized to 60 mg, and addition of placebo to 120 mg dose for those randomized to 120 mg). However, 2/70 patients randomized to 60 mg and then up-titrated to 120 mg after 4 weeks had reduction in MADRS ≥50% after 4 weeks, and 3/64 patients randomized to 120 mg and then given placebo in addition after 4 weeks had reduction in MADRS ≥50% after 4 weeks.
Time Frame: 4 to 8 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- Duloxetine 60 mg Responders: 60mg QD for 8 weeks
- Duloxetine 60 mg Non-Responders: 60mg QD for 4 weeks then 60mg BID for 4 weeks
- Duloxetine 120 mg Responders: 60mg BID for 8 weeks
- Duloxetine 120 mg Non-Responders: 60mg BID for 8 weeks (placebo added at Week 4)
Arm/Group | Duloxetine 60 mg Responders | Duloxetine 60 mg Non-Responders | Duloxetine 120 mg Responders | Duloxetine 120 mg Non-Responders
Number analyzed (Participants) | 96 | 70 | 106 | 64
percentage of participants
  ≥50% Reduction in MADRS Week 4 | 100.0 | 2.9 | 100.0 | 4.7
  ≥50% Reduction in MADRS Week 6 | 94.8 | 52.9 | 98.1 | 39.1
  ≥50% Reduction in MADRS Week 8 | 93.8 | 65.7 | 98.1 | 54.7
  ≥50% Reduction in HAMD-6 Week 4 | 88.5 | 10.0 | 85.8 | 12.5
  ≥50% Reduction in HAMD-6 Week 6 | 90.6 | 47.1 | 90.6 | 31.3
  ≥50% Reduction in HAMD-6 Week 8 | 92.7 | 60.0 | 95.3 | 46.9

10. Secondary Outcome: Patients Reaching Remission
Description: Major Depressive Disorder remission was defined as a total MADRS score ≤12 at Week 8.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine 60 mg Responders | Duloxetine 60 mg Non-Responders | Duloxetine 120 mg Responders | Duloxetine 120 mg Non-Responders
Number analyzed (Participants) | 96 | 70 | 106 | 64
participants
  Remission at Week 8 - Yes | 85 | 29 | 94 | 18
  Remission at Week 8 - No | 11 | 41 | 12 | 46

11. Secondary Outcome: Reason for Living (RFL) Questionnaire Mean Scores at Baseline and Week 8
Description: The RFL questionnaire is an instrument that evaluates patient's reasons for not committing suicide using a 6-point rating scale, where 1 is "not at all important" and 6 is "extremely important". The questionnaire required participants to rate how important each item would be for living, if suicide was contemplated. Mean scores could range from 0 to 6.
Time Frame: Baseline and Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg Responder | Duloxetine 60 mg Non-Responder | Duloxetine 120 mg Responder | Duloxetine 120 mg Non-Responder | Duloxetine 60 mg (All) | Duloxetine 120 mg (All)
Number analyzed (Participants) | 96 | 70 | 106 | 64 | 166 | 170
units on a scale
  Week 0 (Baseline) (n=96, n=66, n=106, n=61) | 4.0 (1.1) | 3.6 (1.0) | 3.7 (1.0) | 3.7 (1.0) | 3.8 (1.1) | 3.7 (1.0)
  Week 8 (n=93, n=63, n=100, n=59) | 4.6 (0.9) | 4.0 (1.2) | 4.6 (0.9) | 3.8 (1.1) | 4.4 (1.1) | 4.3 (1.1)
  Change from Baseline (n=93, n=59, n=100, n=57) | 0.7 (0.9) | 0.4 (0.8) | 0.8 (0.8) | 0.1 (0.9) | 0.6 (0.9) | 0.6 (0.9)
Statistical Analysis 1: Comparison: Duloxetine 60 mg Responder; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value for Change from Baseline (within group); paired t-test
Statistical Analysis 2: Comparison: Duloxetine 60 mg Non-Responder; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — P-value for Change from Baseline (within group); paired t-test
Statistical Analysis 3: Comparison: Duloxetine 120 mg Responder; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — P-value for Change from Baseline (within group); paired t-test
Statistical Analysis 4: Comparison: Duloxetine 120 mg Non-Responder; Test type: Superiority or Other; p = 0.28, t-test, 2 sided — P-value for Change from Baseline (within group); paired t-test

12. Secondary Outcome: Utilization of Allowed Hypnotic and/or Anxiolytic Co-Medication
Description: Number of participants using medication for anxiety and sleep disturbances.
Time Frame: over 8 weeks
Population: All randomized participants who received at least one dose of study drug; had baseline and at least one post-baseline value. Last observation carried forward. The total number of patients with hypnotics and anxiolytics concomitant therapies was 125 (Duloxetine 60mg) and 123 (Duloxetine 120mg).
Measure: Number; unit: participants
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 166 | 170
participants
  Medication Taken Before Start of Study (Week -1) | 65 | 59
  Medication Taken Between Week -1 and Week 0 | 93 | 88
  Medication Taken Between Week 0 and Week 1 | 95 | 89
  Medication Taken Between Week 1 and Week 2 | 80 | 84
  Medication Taken Between Week 2 and Week 3 | 62 | 67
  Medication Taken Between Week 3 and Week 4 | 55 | 58
  Medication Taken Between Week 4 and Week 6 | 47 | 49
  Medication Taken Between Week 6 and Week 8 | 51 | 52
  Medication Taken After Week 8 | 18 | 10
  Medication Not Taken Between Consecutive Visits | 8 | 8

13. Secondary Outcome: Number of Patients With Potentially Clinically Significant Laboratory Findings
Description: Laboratory results that were potentially clinically significant.
Time Frame: over 8 weeks
Population: All randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 167 | 171
participants
  Decreased Haematocrit (n=155, n=159) | 0 | 1
  Decreased Haemoglobin (n=156, n=160) | 2 | 2
  Decreased Red Cell Count (n=156, n=160) | 0 | 1
  Increased Mean Cell Volume (n=155, n=159) | 0 | 1
  Decreased White Cell Count (n=156, n=160) | 1 | 2
  Decreased Sodium (n=160, n=163) | 1 | 0
  Increased Potassium (n=159, n=163) | 0 | 1
  Increased Aspartate Transaminase (n=158, n=161) | 2 | 0
  Increased Alanine Transaminase (n=159, n=161) | 3 | 1
  Increased Alkaline Phosphatase (n=161, n=163) | 0 | 1
  Increased Gamma-Glutamyl Transferase (n=161,n=163) | 2 | 0
  Increased Creatine Kinase (n=159, n=161) | 6 | 3
  Decreased Glucose (n=158, n=162) | 1 | 1
  Increased Cholesterol (n=160, n=163) | 1 | 0
  Increased Total Bilirubin (n=159, n=161) | 0 | 1
  Increased Uric Acid (n=160, n=163) | 0 | 2
  Decreased Albumin (n=158, n=161) | 0 | 1

14. Secondary Outcome: Discontinuations Due to Adverse Events (AE)
Description: Listing of adverse events (AE) that led to treatment discontinuation (DC).
Time Frame: over 8 weeks
Population: All randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 167 | 171
participants
  Total Number of Patients With AEs Leading to DC | 11 | 9
  Suicide Attempt | 3 | 0
  Suicidal Ideation | 2 | 1
  Hypothyroidism | 1 | 0
  Depression | 1 | 2
  Major Depression | 1 | 0
  Psychotic Disorder | 1 | 0
  Schizoaffective Disorder | 1 | 0
  Self-Injurious Behaviour | 1 | 0
  Headache | 1 | 0
  Nausea | 1 | 0
  Irritability | 1 | 0
  Brain Neoplasm | 0 | 1
  Dizziness | 0 | 1
  Sedation | 0 | 1
  Serotonin Syndrome | 0 | 1
  Upper Abdominal Pain | 0 | 1
  Drug Eruption | 0 | 1
  Renal Failure | 0 | 1
  Urinary Retention | 0 | 1

15. Secondary Outcome: Number of Participants Experiencing High Values for Vital Signs at Any Time During the Study
Description: Systolic and diastolic blood pressure and pulse rate were measured after 2 minutes rest in a supine position. High values were: diastolic blood pressure ≥90 mm Hg and increase from baseline of ≥10 mm Hg; systolic blood pressure ≥140 mm Hg and increase from baseline of ≥10 mm Hg; pulse rate ≥100 beats per minute (bpm) and an increase of ≥10 bpm from baseline.
Time Frame: over 8 weeks
Population: All randomized participants with at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 167 | 171
participants
  High Systolic Blood Pressure | 23 | 25
  High Diastolic Blood Pressure | 28 | 37
  High Pulse Rate | 10 | 14

16. Secondary Outcome: Change From Baseline to Week 4 and Week 8 in Weight
Description: Change in weight = Post-baseline visit minus baseline.
Time Frame: Baseline to Weeks 4 and 8
Population: All randomized participants with at least one dose of study drug and a baseline and at least one post-baseline value. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Number analyzed (Participants) | 167 | 171
kilograms
  Change from Baseline to Week 4 (n=163,n=167) | 0.1 (2.0) | 0.0 (2.3)
  Change from Baseline to Week 8 (n=163, n=168) | 0.5 (2.9) | 0.1 (2.8)

ADVERSE EVENTS:
Arm/Group | Duloxetine (60 mg) | Duloxetine (120 mg)
Serious Adverse Events (participants affected / at risk) | 7 | 6
Other Adverse Events (participants affected / at risk) | 95 | 85
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine (60 mg) | Duloxetine (120 mg)
Irritability (General disorders) | 1/167 (1) | 0/171 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/167 (1) | 0/171 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/167 (0) | 1/171 (1)
Serotonin syndrome (Nervous system disorders) | 0/167 (0) | 1/171 (1)
Anxiety (Psychiatric disorders) | 0/167 (0) | 2/171 (2)
Depression (Psychiatric disorders) | 0/167 (0) | 2/171 (2)
Self injurious behaviour (Psychiatric disorders) | 1/167 (1) | 0/171 (0)
Suicidal ideation (Psychiatric disorders) | 3/167 (3) | 0/171 (0)
Suicide attempt (Psychiatric disorders) | 4/167 (4) | 0/171 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Duloxetine (60 mg) | Duloxetine (120 mg)
Constipation (Gastrointestinal disorders) | 8/167 (8) | 16/171 (21)
Diarrhoea (Gastrointestinal disorders) | 7/167 (7) | 4/171 (4)
Dry mouth (Gastrointestinal disorders) | 8/167 (8) | 12/171 (14)
Nausea (Gastrointestinal disorders) | 37/167 (42) | 21/171 (25)
Nasopharyngitis (Infections and infestations) | 4/167 (6) | 9/171 (9)
Headache (Nervous system disorders) | 26/167 (37) | 19/171 (19)
Tremor (Nervous system disorders) | 3/167 (3) | 8/171 (8)
Insomnia (Psychiatric disorders) | 4/167 (8) | 7/171 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9/167 (9) | 5/171 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days